CLINICAL TRIAL: NCT00984113
Title: An Open-label, Parallel-group Study to Determine the Single and Multiple Dose Pharmacokinetics of Elinogrel and Its Metabolite in Patients With Mild, Moderate, and Severe Renal Impairment Compared to Healthy Subjects
Brief Title: Pharmacokinetics of Elinogrel in Healthy Volunteers and Patients With Mild, Moderate, and Severe Renal Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: For administrative reasons. Enrollment was sufficient to have statistical power without compromising the integrity of the study data
Sponsor: Portola Pharmaceuticals (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Matthew W. McClure, MD, Portola Pharmaceuticals, Inc.
Organization: Alexion Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-115 / CPRT128A2104
Record Dates: First submitted 2009-09-16; First posted 2009-09-25 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Renal Impairment
Keywords: Elinogrel; Renal impairment; Healthy; Kidney dysfunction
MeSH Terms: conditions — Renal Insufficiency | interventions — elinogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- A-Patients with mild renal impairment (Experimental)
  Interventions: Drug: Elinogrel
- B-Healthy subjects matched to Group A (Experimental)
  Interventions: Drug: Elinogrel
- C-Patients with moderate renal impairment (Experimental)
  Interventions: Drug: Elinogrel
- D-Healthy subjects matched to Group C (Experimental)
  Interventions: Drug: Elinogrel
- E-Patients with severe renal impairment (Experimental)
  Interventions: Drug: Elinogrel
- F-Healthy subjects matched to Group E (Experimental)
  Interventions: Drug: Elinogrel

INTERVENTIONS:
Drug: Elinogrel — 100 mg elinogrel b.i.d. with aspirin q.d. for 7 days and aspirin alone for 4 days (Dose of aspirin is 81 mg in the US and 100 mg in Germany)
  Other Names: PRT060128

SUMMARY:
The purpose of the study is to determine the pharmacokinetics and safety of elinogrel and its metabolite in patients with mild, moderate, and severe renal impairment compared to healthy volunteers.

DETAILED DESCRIPTION:
Multiple-dose, open-label parallel-group design in patients with mild, moderate or severe renal impairment and age (±7 years), sex and weight (±15% BMI) matched healthy subjects.

* mild renal impairment: CrCl from 50 to ≤80 ml/min
* moderate renal impairment: CrCl from 30 to <50 ml/min
* severe renal impairment: CrCl of <30 ml/min

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and sign the written informed consent
* Subjects should have either normal renal function or have stable renal disease

Exclusion Criteria:

* History of heart disease
* Unstable or clinically significant other disorders such as respiratory, hepatic, metabolic, psychiatric or gastrointestinal disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of elinogrel and its metabolite | 7 days
  The PK parameters calculated for both elinogrel and PRT060301 were:
  * AUC0-12h, Cmax, and Tmax on Day 1/Day 7 and T1/2, RACC & CLR on Day 7
  * For elinogrel only, CLss/F and Vss/F were also calculated

SECONDARY OUTCOMES:
Safety assessments will include vital signs, electrocardiograms and adverse events | 9 days
  Safety assessments consisted of collecting all adverse events (AEs), serious adverse events (SAEs), with their severity and relationship to study drug, and pregnancies, regular monitoring of hematology, blood chemistry and urinalysis performed at study center. Safety assessments also included periodic ECG evaluations, assessments of vital signs, physical condition, and body weight.
Measures of platelet function | 7 days
  Platelet aggregation using VerifyNOW P2Y12 assay and thrombi formation using Portola's proprietary PCA (Perfusion Chamber Assay).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W McClure, MD, Study Director — Portola Pharmaceuticals Inc.
Locations (2):
- United States (2):
  - DaVita Clinical Research, Minneapolis, Minnesota
  - NOCR-Knoxville, Knoxville, Tennessee